CLINICAL TRIAL: NCT04857918
Title: The UBC Socializing Together While Running InDEpendently (STRIDE) Pilot Trial: A Social Identity Informed Virtual Running Group Program
Brief Title: Assessing the Feasibility and Acceptability of a Social Identity Informed Virtual Running Group Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Social Sciences and Humanities Research Council of Canada (Other); University of Victoria (Other)
Responsible Party: Principal Investigator, Mark Beauchamp, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H20-03151
Record Dates: First submitted 2021-04-12; First posted 2021-04-23 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Well-being; Physical Activity; Identity, Social
Keywords: Feasibility; Acceptability; Well-being; Social identity; Exercise identity; Exercise; Physical Activity; Social Support
MeSH Terms: conditions — Motor Activity; Social Identification

STUDY DESIGN:
Intervention Model Description: The study will utilize a two-arm, parallel group, unblinded randomized controlled pilot trial design. UBC undergraduate students (N = 60) will be equally randomized to either an eight-week social identity building virtual running group (n = 30) or an eight-week control group (n = 30).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social identity informed virtual running group (Experimental): Participants will join running groups of six people (males and females) for eight weeks. Each running group will be given the group goal/challenge to collectively run/brisk walk the distance across the province of British Columbia (940 km) over the course of the eight week intervention (Estabrooks et al., 2008), and encouraged to complete 150 minutes of moderate-to-vigorous exercise per week. Participants can record other moderate-to-vigorous exercise to contribute to the group goal. Running groups will be created on the fitness application Strava, and participants will record/post their runs on the Strava app so that members of their running group can provide 'kudos' and words of encouragement. Running groups will have a weekly a coffee chat (via Zoom) to socialize and discuss their experiences running/exercising and progress and challenges associated with meeting the group goal. Participants will also be provided running tip videos, phone armbands, and t-shirts with the study logo.
  Interventions: Behavioral: Virtual running group program
- Attention control group (Active Comparator): This group of participants will act as an attention control condition. This group will be asked to download the fitness application Strava to their smartphone, and track all of their runs and walks on Strava. Similar to the intervention group, participants will be provided with phone armbands to carry their phone during a run or walk so they can record the run or walk on Strava, and will be asked to try participating in 150 minutes of moderate-to-vigorous exercise per week.
  Interventions: Behavioral: Attention Control: Fitness Application Strava

INTERVENTIONS:
Behavioral: Virtual running group program — The intervention will include an eight-week virtual running group program hosted on online platforms such as Zoom and the fitness application Strava. Participants will be placed in running groups of 6 people, and each running group will have the collective goal to run/walk the distance across the province of B.C., (940 km) and will meet weekly over Zoom to socialize and discuss running topics and their progress towards the group goal. Participants will receive a t-shirt with the STRIDE logo and a phone armband for carrying their smart phone during runs and walks.
  Arms: Social identity informed virtual running group
Behavioral: Attention Control: Fitness Application Strava — The attention control condition will be instructed to record their exercise using the Strava application, and will be encouraged to participate in 150 minutes of moderate-to-vigorous exercise each week of the intervention.
  Arms: Attention control group

SUMMARY:
The STRIDE Pilot Trial is a randomized controlled pilot trial that will utilize social identity informed virtual running groups to support underactive undergraduate students' well-being and exercise behaviour. The main outcomes of this study are to determine whether the intervention is feasible and acceptable to conduct as a full-scale efficacy trial. Secondary outcomes of interest include changes in participants' exercise identity, exercise behaviour, perceived social support, and well-being. Participants' perceived social identification with their running group will also be assessed at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* currently residing in Canada
* age 18+
* enrolled in undergraduate studies at the University of British Columbia
* underactive (i.e., currently participating in less than the Canadian physical activity guidelines of 150 minutes of physical activity per week)
* not experience any health contraindication which might prevent that person from participating in moderate-to-vigorous intensity exercise.
* able to speak and read English
* own a smart phone
* have home access to the internet and a device with camera functionality

Exclusion Criteria:

* If a potential participant has a medical contraindication (flagged through the PAR-Q+ and ePARmedX) and have NOT been cleared to participate in physical activity by their physician they are then ineligible to participate in the study
* Participants are asked to record their running and walking behaviour on the fitness application Strava, and participate in Zoom coffee chats with their running group. If an individual is unwilling to download the Strava application and/or do not want to use Zoom they will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Feasibility and Acceptability: Participant interest in the program | Recorded from recruitment to follow-up (Week 8)
  Total number of individuals expressing interest in the program.
Feasibility and Acceptability: Participant enrolment | Follow up (Week 8)
  Participant enrolment will be assessed with the total number of participants enrolled in the study.
Feasibility and Acceptability: Affective attitudes towards exercise | Change from Baseline (Week 0) to follow-up (Week 8)
  Participants' affective attitudes towards exercise will be assessed using four bipolar semantic differential adjectives (Conner et al., 2011) rated on a seven-point scale ranging from 1 to 7 (pleasant-unpleasant; enjoyable-unenjoyable; exciting-boring; satisfying-unsatisfying). The four items will be mean-scored (potential range 1-7), with higher scores reflecting higher positive affective attitudes towards exercise, and a more positive outcome.
Feasibility and Acceptability: Program satisfaction | Follow-up (Week 8)
  One item, adapted from a pilot study conducted by Vincze et al. (2018), will be used to assess general satisfaction with the program. Participants (virtual running program only) will rate their satisfaction with the STRIDE program on a 5-point Likert-type scale anchored by 1 (Not at all satisfied) to 5 (Extremely satisfied). Higher scores will reflect greater program satisfaction and a more positive outcome.
Feasibility and Acceptability: Study Retention | Recorded from Baseline (Week 0) to follow up (Week 8)
  The percentage of participants who adhere to the study.
Feasibility and Acceptability: Questionnaire completion rates | Recorded from Baseline (Week 0) to follow up (Week 8)
  Percentage of questionnaires completed.
Feasibility and Acceptability: Program attendance | Recorded from Baseline (Week 0) to follow up (Week 8)
  Percentage of weekly Zoom meetings attended.
Feasibility and Acceptability: Semi structured interviews | Follow up (Week 8)
  10 semi-structured interviews will be conducted with members of the intervention group to assess participants' experiences and satisfaction with the program, as well as their perceptions of social support, group identification, and exercise identity throughout the program.

SECONDARY OUTCOMES:
Well-Being (Psychological Flourishing) | Change from Baseline (Week 0) to follow-up (Week 8)
  Domain general well-being will be assessed using the 8-item Flourishing Scale from Diener et el., (2010). Participants will respond to the 8 flourishing items on a 7-point Likert-type scale anchored by 1 (Strongly disagree) to 7 (Strongly agree). The 8 items will be mean-scored (potential range 1-7), with higher scores indicating higher psychological flourishing and a more positive outcome.
Perceived Social Support Received in the Context of Exercise | Change from Baseline (Week 0) to follow-up (Week 8)
  Social support in the context of exercise will be assessed using a four-item social support scale (Gleibs et al., 2011; Haslam et al., 2005) adapted for the context of exercise participation. Participants will respond to the 4 social support items on a 5-point Likert-type scale anchored by 1 (Strongly Disagree) to 5 (Strongly Agree). The 4 items will be mean-scored (potential range 1-5), with higher scores reflecting greater perceived social support from others in the context of exercise and a more positive outcome.
Well-Being (Subjective Vitality) | Change from Baseline (Week 0) to follow-up (Week 8)
  Participants will complete the six-item (Bostic et al., 2000) Subjective Vitality Scale (SVS; Ryan & Frederick, 1997) adapted for the context of exercise behaviour. Participants will respond to the 6 exercise-related subjective vitality items on a 7-point Likert-type scale anchored by 1 (Not at All True) to 7 (Very True). The 6 items will be mean-scored (potential range 1-7), with higher scores reflecting greater subjective experiences of vitality in the context of exercise and a more positive outcome.
Exercise Identity | Change from Baseline (Week 0) to follow-up (Week 8)
  Participants will complete the nine-item Exercise Identity Scale (Anderson & Cychosz, 1994). Participants will respond to the 9 exercise identity items on a 7-point Likert-type scale anchored by 1 (Strongly Disagree) to 7 (Strongly Agree). Consistent with Wilson and Muon (2008), two separate scores will be calculated to reflect the role-identity dimension and the exercise beliefs dimension of the scale. Items 1, 2, and 6 will be mean-scored (potential range 1-7), with higher score reflecting a greater role identity in relation to exercise behaviour, and items 3, 4, 5, 7, 8, and 9 will be mean-scored (potential range 1-7), with higher scores reflecting greater exercise-related beliefs and a more positive outcome.
Social Identification with the Running Group | Follow-up (Week 8)
  Using a four-item social identification scale (Doosje et al., 1995), participants in the intervention condition will respond to four items inquiring the degree to which they positively identify with their running group. Participants will respond to the 4 social identification items using a 7-point Likert-type scale anchored by 1 (Strongly Disagree) to 7 (Strongly Agree). The 4 items will be mean-scored (potential range 1-7), with higher scores reflecting stronger positive identification with the running group and a more positive outcome.
Exercise Behaviour | Change from Baseline (Week 0) to follow-up (Week 8)
  In reference to the past month, participants will report the number of times per week (on average) they engaged in mild, moderate, and vigorous exercise using the Godin Leisure Time Exercise Questionnaire (Godin & Shephard, 1985), and the average duration of mild, moderate, and vigorous exercise sessions (Courneya et al., 2004). Consistent with Courneya et al. (2004), the researchers will create an indicator of average weekly moderate-to-vigorous exercise minutes (in past month) for each participant using the following equation: (number of moderate exercise bouts x average minutes per bout) + (number of vigorous exercise bouts x average minutes per bout). The scores will have a minimum value of 0 minutes, with more minutes indicating greater participation in moderate-to-vigorous exercise and a more positive outcome.
Weekly exercise behaviour (activity type) | Week 1, 2, 3, 4, 5, 6, 7, and 8
  Participants will log their daily exercise (type of activity) at the end of each week
Weekly exercise behaviour (activity duration) | Week 1, 2, 3, 4, 5, 6, 7, and 8
  Participants will log their daily exercise (duration of activity) at the end of each week
Demographics | Baseline (Week 0)
  Items addressing sex/gender, age, ethnicity, height, weight, residence (City, Province), disability, marital status, swelling type, living situation (alone, others), undergraduate major

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Anderson DF, Cychosz CM. Development of an exercise identity scale. Percept Mot Skills. 1994 Jun;78(3 Pt 1):747-51. doi: 10.1177/003151259407800313. PMID 8084685
- [Background] Bostic, T. J., Rubio, D. M., & Hood, M. (2000). A validation of the subjective vitality scale using structural equation modelling. Social Indicators Research, 52(3), 313-324. https://doi.org/10.1111/j.1541-0072.1977.tb01338.x
- [Background] Conner M, Rhodes RE, Morris B, McEachan R, Lawton R. Changing exercise through targeting affective or cognitive attitudes. Psychol Health. 2011 Feb;26(2):133-49. doi: 10.1080/08870446.2011.531570. PMID 21318926
- [Background] Courneya KS, Jones LW, Rhodes RE, Blanchard CM. Effects of different combinations of intensity categories on self-reported exercise. Res Q Exerc Sport. 2004 Dec;75(4):429-33. doi: 10.1080/02701367.2004.10609176. No abstract available. PMID 15673042
- [Background] Diener, E., Wirtz, D., Tov, W., Kim-Prieto, C., Choi, D.-W., Oishi, S., & Biswas-Diener, R. (2010). New well-being measures: Short scales to assess flourishing and positive and negative feelings. Social Indicators Research, 97(2), 143-156.
- [Background] Doosje, B., Ellemers, N., Spears, R. (1995) Perceived intragroup variability as a function of group status and identification. Journal of Experimental Social Psychology 31(5): 410-436.
- [Background] Estabrooks PA, Bradshaw M, Dzewaltowski DA, Smith-Ray RL. Determining the impact of Walk Kansas: applying a team-building approach to community physical activity promotion. Ann Behav Med. 2008 Aug;36(1):1-12. doi: 10.1007/s12160-008-9040-0. Epub 2008 Jul 8. PMID 18607666
- [Background] Gleibs IH, Haslam C, Haslam SA, Jones JM. Water clubs in residential care: is it the water or the club that enhances health and well-being? Psychol Health. 2011 Oct;26(10):1361-77. doi: 10.1080/08870446.2010.529140. Epub 2011 May 23. PMID 21598183
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Haslam SA, O'Brien A, Jetten J, Vormedal K, Penna S. Taking the strain: social identity, social support, and the experience of stress. Br J Soc Psychol. 2005 Sep;44(Pt 3):355-70. doi: 10.1348/014466605X37468. PMID 16238844
- [Background] Ryan RM, Frederick C. On energy, personality, and health: subjective vitality as a dynamic reflection of well-being. J Pers. 1997 Sep;65(3):529-65. doi: 10.1111/j.1467-6494.1997.tb00326.x. PMID 9327588
- [Background] Vincze L, Rollo ME, Hutchesson MJ, Callister R, Collins CE. VITAL change for mums: a feasibility study investigating tailored nutrition and exercise care delivered by video-consultations for women 3-12 months postpartum. J Hum Nutr Diet. 2018 Jun;31(3):337-348. doi: 10.1111/jhn.12549. Epub 2018 Mar 15. PMID 29543356
- [Background] Wilson, P. M., & Muon, S. (2008). Psychometric properties of the exercise identity scale in a university sample. International Journal of Sport and Exercise Psychology, 6, 115-131.
- [Derived] Wierts CM, Rhodes RE, Faulkner G, Zumbo BD, Beauchamp MR. An online delivered running and walking group program to support low-active post-secondary students' well-being and exercise behavior during the COVID-19 pandemic: a pilot randomized controlled trial. J Behav Med. 2024 Dec;47(6):935-950. doi: 10.1007/s10865-024-00516-z. Epub 2024 Sep 3. PMID 39225842

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT04857918/Prot_SAP_001.pdf